CLINICAL TRIAL: NCT00809809
Title: A Randomized, Double-blind, Placebo-controlled, Multi-Center Trial of Zinc for the Treatment of Herpes Simplex Labialis (HSL)
Brief Title: Zinc for the Treatment of Herpes Simplex Labialis (HSL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Integrative Medicine Institute (Other)
Collaborators: Women's Health Services, Santa Fe, New Mexico (Other); Southwest College of Naturopathic Medicine (Other); Beth Israel Medical Center (Other); Matrixx Initiatives, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMIZnc2008
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2013-11

CONDITIONS: Herpes Simplex Labialis
Keywords: Cold sores; Zinc; HSL; Herpes simple labialis
MeSH Terms: conditions — Herpes Labialis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zinc gluconate (Active Comparator): Oral swabs containing homeopathic Zinc gluconate
  Interventions: Drug: Zicam (Ionic zinc)
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Zicam (Ionic zinc) — 33mmol/l of ionic zinc
  Other Names: Homeopathic Zinc gluconate
  Arms: Zinc gluconate
Drug: placebo — placebo swab
  Other Names: placebo swab
  Arms: Placebo

SUMMARY:
Evaluate the effectiveness of a topical preparation of zinc to treat cold sores.

DETAILED DESCRIPTION:
Zinc salts irreversibly inhibit herpes virus replication in vitro and are effective in treating herpes infections in vivo and have been shown in a clinical trial to be a effective topical treatment for HSL. Zinc salt solutions applied to herpetic lesions decrease viral load and markedly improve healing rates, relieving the symptoms of herpes as healing occurs. Zinc swabs contain 33 mmol/l of ionic Zinc in an emulsification of Benzalkonium chloride, glycerin, hydroxyethylcellulose, sodium chloride, and sodium hydroxide (ph 7.2). Zinc gluconate is monographed in the Homeopathic Pharmacopoeia of the United States (HPUS) and one of OTC indications for Zinc and its salts is for the treatment of cold sores.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of HSL with at least 2 episodes/year for the past two years that have proceeded beyond the prodromal (initial) stage
* Male or female subjects between 18 and 65 years of age
* Symptoms or signs of HSL for less than one day (max. 36 hours from onset of symptoms to first visit)
* Confirmation of HSL by a clinician at the study site
* Willing to comply with study instructions and sign an informed consent

Exclusion Criteria:

* HSL symptoms or signs for more than one day
* Cold sore outbreak within the past 2 weeks
* Previous participation in this clinical trial
* Topical or oral antiviral drug use in the past 1 week
* Immune deficiency (HIV positive), chronic steroid therapy, present anti-neoplastic or radiation therapy, Hodgkin's disease, splenectomy, leukemia, myeloma, lymphoma, or another condition/drug per judgment of attending health care professional) or currently taking immune suppressive drugs. Previous organ or bone marrow transplant.
* Pregnancy or lactation
* Unable to travel to the clinic area for the required visits
* Apparent inability to understand or follow the instructions associated with the clinical study
* History of adverse events to the study material or facial cosmetics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Riley, MD, Principal Investigator — University of New Mexico
Locations (3):
- United States (3):
  - Steven Messer ND, DHANP, Tempe, Arizona
  - Deborah Thompson, MD MSPH, Santa Fe, New Mexico
  - Benjamin Kligler, MD, New York, New York

REFERENCES:
- [Background] Godfrey HR, Godfrey NJ, Godfrey JC, Riley D. A randomized clinical trial on the treatment of oral herpes with topical zinc oxide/glycine. Altern Ther Health Med. 2001 May-Jun;7(3):49-56. PMID 11347285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 3 medical clinics: Women's Health Services, Santa Fe, NM; Continuum Center, NYC, NY; SCNM medical Clinic, Scottsdale, Az
Pre-assignment Details: Subjects were excluded if they had HSL for more than one day
Groups:
- Active Treatment: Active medication - Zinc Swabs
- Placebo Treatment: Placebo medication - Swabs identical to medication group
Period: Overall Study
Arm/Group | Active Treatment | Placebo Treatment
Started | 78 | 79
Completed | 75 (3 dropped from the study when it was discovered they met the exclusion criteria) | 77 (2 dropped from the study when it was discovered they met the exclusion criteria)
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo Treatment | Total
Number analyzed (Participants) | 78 | 79 | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 79 | 157
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (11.8) | 43.8 (12.5) | 43.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 62 | 122
  Male | 18 | 17 | 35
Region of Enrollment [Number; unit: participants]
  United States | 78 | 79 | 157

OUTCOME MEASURES:

1. Primary Outcome: Zicam Was Compared to Placebo as a Treatment of Recurrent HSL From the Date and Time of the Initiation of Therapy Until the Date and Time of Resolution of the Lesion or After 14 Days of Treatment, Whichever Comes First.
Description: Zinc gluconate swabs were compared as a treatment of recurrent HSL compared to placebo from the date and time of the initiation of therapy until the date and time of resolution of the lesion or after 14 days of treatment, whichever comes first.
Time Frame: 14 days
Population: 5 subjects met exclusion criteria and were excluded from analysis. 2 subjects used concomitant medications and were excluded from the final analysis. Twelve subjects with recurrent HSL enrolled twice, only the 1st enrollment was included in the analysis. 2 subjects had family enroll who were excluded from analysis. Analysis - 134 subjects.
Measure: Median (95% Confidence Interval); unit: Days to resolution
Arm/Group | Active Treatment | Placebo Treatment
Number analyzed (Participants) | 61 | 73
Days to resolution | 8 [0 to 16] | 6 [0 to 21]

2. Secondary Outcome: Compare Zicam to Placebo on the Incidence of, Speed of, and the Rate of Healing for Aborted Cold Sore Lesions.
Time Frame: 14 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14 days per subject
Arm/Group | Active Treatment | Placebo Treatment
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/79
Other Adverse Events (participants affected / at risk) | 0/78 | 0/79

LIMITATIONS AND CAVEATS:
There may have been differences between the populations in the different study sites that influenced the outcome of this clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No